CLINICAL TRIAL: NCT00004285
Title: Randomized Study of Standard vs High Amount of Hemodialysis Using Low vs High Flux Dialyzer Membranes for End Stage Renal Disease
Brief Title: Effect of Dialysis Dose and Membrane Flux in Maintenance Hemodialysis
Acronym: HEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Rochester (Other); The Cleveland Clinic (Other); Tufts Medical Center (Other); Vanderbilt University (Other); Icahn School of Medicine at Mount Sinai (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Washington University School of Medicine (Other); University of Illinois at Chicago (Other); Main Line Health (Other); Emory University (Other); Duke University (Other); University of Texas Southwestern Medical Center (Other); Brigham and Women's Hospital (Other); Wake Forest University Health Sciences (Other); University of Utah (Other); University of California, Davis (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 199/11704; U01DK046109 (NIH); U01DK046114 (NIH); U01DK046126 (NIH); U01DK046140 (NIH); U01DK046143 (NIH); U01DK049240 (NIH); U01DK049241 (NIH); U01DK049242 (NIH); U01DK049243 (NIH); U01DK049244 (NIH); U01DK049249 (NIH); U01DK049252 (NIH); U01DK049254 (NIH); U01DK049259 (NIH); U01DK049261 (NIH); U01DK049264 (NIH); U01DK049271 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Kidney Failure, Chronic; Rare Diseases; Urogenital Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Standard dose, low flux hemodialysis (Active Comparator)
  Interventions: Device: Standard dose, low flux hemodialysis
- Standard dose, high flux hemodialysis (Experimental)
  Interventions: Device: Standard dose, high flux hemodialysis
- High dose, low flux hemodialysis (Experimental)
  Interventions: Device: High dose, low flux hemodialysis
- High dose, high flux hemodialysis (Experimental)
  Interventions: Device: High dose, high flux hemodialysis

INTERVENTIONS:
Device: Standard dose, low flux hemodialysis
  Arms: Standard dose, low flux hemodialysis
Device: Standard dose, high flux hemodialysis
  Arms: Standard dose, high flux hemodialysis
Device: High dose, low flux hemodialysis
  Arms: High dose, low flux hemodialysis
Device: High dose, high flux hemodialysis
  Arms: High dose, high flux hemodialysis

SUMMARY:
OBJECTIVES: I. Evaluate whether hemodialysis providing a 2-pool, variable volume urea kinetic modelling value of 1.05 versus 1.45 reduces mortality and morbidity in patients with end stage renal disease.

II. Compare the efficacy of high versus low flux dialyzer membranes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, age, and diabetes prior to dialysis initiation.

Patients are randomly assigned to 1 of 4 groups: moderate dose dialysis, low flux membrane; high dose dialysis, low flux membrane; moderate dose dialysis, high flux membrane; or high dose dialysis, high flux membrane. Moderate dose is a target eKt/V of 1.05 and high dose is 1.45. The dose and delivery of dialysis are measured monthly by the equilibrated fractional clearance of urea (eKt/V) calculated with double pool kinetics.

Patients are dialyzed 3 times a week in the shortest possible time (minimum 2.5 hours), adjusted for adequate fluid removal. General medical care, protein and calorie intake, and dialyzer reuse and other aspects of dialysis therapy are standardized. The protocol document lists approved dialyzers; no unsubstituted cellulosic membranes are permitted.

The intervention phase of this study is 5 years. Patients are followed for survival.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* End stage renal disease that requires in-center hemodialysis 3 times/week On hemodialysis for at least 3 months (6 months following renal transplant)
* No scheduled renal transplant from living donor

--Prior/Concurrent Therapy--

* No concurrent intervention studies unless ancillary to this protocol No concurrent investigational drugs

--Patient Characteristics--

* Hepatic: Albumin at least 2.6 g/dL by nephelometry No cirrhosis with encephalopathy or abnormal PT
* Renal: Urea clearance (interdialytic) no greater than 1.5 mL/min per 35 liters total urea volume
* Cardiovascular: No New York Heart Association class IV congestive heart failure despite maximal therapy No unstable angina No new onset angina No recent exacerbation of frequency, duration, or severity of angina
* Pulmonary: No chronic pulmonary disease requiring supplemental oxygen
* Other: Not hospitalized in acute or long term care facility at entry No active malignancy requiring chemotherapy or radiotherapy No AIDS No active systemic infection, e.g., tuberculosis or fungal infection No mental incompetence or other contraindication to protocol therapy Not pregnant Geographically available for treatment at participating institution No more than 20 missed treatments/year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1846 (Actual)
Dates: Start 1995-03 (Actual); Primary Completion 2001-12-31 (Actual); Study Completion 2001-12-31 (Actual)

PRIMARY OUTCOMES:
Death from any cause | 5 years

SECONDARY OUTCOMES:
First hospitalization for cardiac causes or death from any cause | 5 years
First hospitalization for infection or death from any cause | 5 years
First >15% decrease in albumin or death from any cause | 5 years
All hospitalizations not related to vascular access | 5 years
Death due to cardiac causes | 5 years
First hospitalization or death due to cardiac causes | 5 years
Death due to infection | 5 years
First hospitalization or death due to infection | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Ornt, Study Chair — University of Rochester
Locations (1):
- University of Rochester School of Medicine, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and samples are available at the NIDDK central repository
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Available since 2009
URL: https://www.niddkrepository.org/studies/hemo/?query=hemo

REFERENCES:
- [Background] Greene T, Beck GJ, Gassman JJ, Gotch FA, Kusek JW, Levey AS, Levin NW, Schulman G, Eknoyan G. Design and statistical issues of the hemodialysis (HEMO) study. Control Clin Trials. 2000 Oct;21(5):502-25. doi: 10.1016/s0197-2456(00)00062-3. PMID 11018567
- [Result] Eknoyan G, Beck GJ, Cheung AK, Daugirdas JT, Greene T, Kusek JW, Allon M, Bailey J, Delmez JA, Depner TA, Dwyer JT, Levey AS, Levin NW, Milford E, Ornt DB, Rocco MV, Schulman G, Schwab SJ, Teehan BP, Toto R; Hemodialysis (HEMO) Study Group. Effect of dialysis dose and membrane flux in maintenance hemodialysis. N Engl J Med. 2002 Dec 19;347(25):2010-9. doi: 10.1056/NEJMoa021583. PMID 12490682